CLINICAL TRIAL: NCT05380076
Title: Effects of Mindfulness, Mobilization of Inner Resources, or Cardiac Biofeedback on Psychophysiological Anticipatory Stress Before OSCE of Medical Students
Brief Title: Effects of Mindfulness, Mobilization of Resources, or Biofeedback on Stress Before OSCE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Claude Bernard University (Other)
Responsible Party: Principal Investigator, Lilot Marc, Principal investigator, Claude Bernard University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: OsceStress
Record Dates: First submitted 2022-05-13; First posted 2022-05-18 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Exam Stress; Stress, Psychological; Stress, Physiological
MeSH Terms: conditions — Stress, Psychological | interventions — Mindfulness; Biofeedback, Psychology

STUDY DESIGN:
Intervention Model Description: 4 parallel groups
Who Masked: Investigator, Outcomes Assessor
Masking Description: Interventions are standardized video tape. Information collected through standardized informatic questionnaires for blinded investigators.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Mindfulness (Experimental): Mindfulness meditation video before the circuit
  Interventions: Other: Mindfulness meditation
- Mobilization of inner resources (Experimental): Standardised video before the circuit
  Interventions: Other: Mobilization of inner resources
- Biofeedback (Experimental): Cardiac biofeedback before the circuit
  Interventions: Other: Biofeedback
- Control (Sham Comparator): Standardised video before the circuit
  Interventions: Other: Mindfulness meditation; Other: Mobilization of inner resources; Other: Biofeedback

INTERVENTIONS:
Other: Mindfulness meditation — 6 minutes of watching a video tape made for the study that inspire mindfulness like meditation just before entering the examination circuit.
  Arms: Control; Mindfulness
Other: Mobilization of inner resources — 6 minutes of watching a video tape made for the study that provide psychological stimulation just before entering the examination circuit
  Arms: Control; Mobilization of inner resources
Other: Biofeedback — 6 minutes of relaxing breathing exercise coupled with heart rate variability biofeedback guided on eMWave Pro software on a computer just before entering the examination circuit.
  Arms: Biofeedback; Control

SUMMARY:
Stress generated during the curriculum might have deleterious effects on the wellbeing and the health of medical students. Objective and Structured Clinical Examinations (OSCEs) will be incorporated soon in the certification process as a final national undergraduate ranking examination. This exam will be an additional major stressor for medical students.

Stress coping strategies could be implemented to help them better prepare for this examination. The aim of this study was to compare the efficiency on stress reduction of three different 6-minutes coping interventions in medical student, few minutes prior to the OSCE.

DETAILED DESCRIPTION:
This randomized, controlled and monocentric study will be conducted during the OSCE tests contributing towards the final exam grades for 4th year medicine students at the Claude Bernard Lyon 1 university.All the students will receive information for the study and sign consent before being randomized into four interventions groups. All the interventions will last six minutes long.

The randomisation groups are:

* Mindfulness through watching/listening video tape
* Mobilization of inner resources through watching/listening video tape
* Cardiac biofeedback guided standardized timing for respiratory rate and with immediate feedback on cardiac variability score
* Unemotional video tape as controlled group

Psychological stress will be measured using short questionnaires and self-rated Visual Analogue Scale (from 0 to 100mm) regarding perceived stress, answered by students before and after intervention. For measuring physiological stress, all the student will be equipped with emWAve® devices that allows us to record heart rate variability during the time of intervention. Students will also answer a questionnaire of personality.

Main objective is to show that interventions are better than control to reduce stress level before OSCE.

The main outcome is to compare the effect of the interventions on physiological stress, using HRV as physiological stress marker.

Secondary outcomes are to compare the effects of the interventions on psychological stress and to compare the specified aspect of the intervention. Finally, our project will permit to assess if the personality modulates the effectiveness of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Adult person
* Registered as medical student at the university
* Participating at OSCE examination
* Have signed an informed consent form.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 490 (Actual)
Dates: Start 2022-05-17 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2023-12-30 (Actual)

PRIMARY OUTCOMES:
Differences of physiological stress | During the 6min long intervention
  Heart rate variability collected by an ear pulse sensor (emWave® device)

SECONDARY OUTCOMES:
Characterisation of the influence of the intervention on Psychological stress | measured two times: just 30 seconds before and after the intervention
  Numerical Visual analog scales (100mm-VAS) on perceived stress (from zero to 100: maximum)
Characterisation of the influence of the intervention on level of inner resources | measured two times: just 30 seconds before and after the intervention
  Numerical 100mm-VAS on level of resourcefulness perceived (from zero to 100: maximum)
Characterisation of the influence of the intervention on self-confidence | measured two times: just 30 seconds before and after the intervention
  Numerical 100mm-VAS on self confidence perceived (from zero to 100: maximum)
Characterisation of intervention on Psychological stress consequences | measured two times: just 1 minute before and after the intervention
  Activation-Deactivation Adjective Check List: for the four subscales (Tension , Calmness, Activation, Deactivation).
Feelings about the intervention | just 2 minutes after the intervention
  Likert Scale assessing feelings about the intervention: Pleasure, Interest, Enthusiasm, Boredom, Frustration, Discouragement, Fun) on a 5 items answers (from not feeling at all, to very importante intensity)
Determining influence of personality traits on the efficiency on the intervention | just 5 minutes after the intervention
  Personality questionnaire (Big-5, 10 items) allowing score in 5 factors of personality (Openness, Consciousness, Extraversion, Agreeableness, Nevrosism).

CONTACTS AND LOCATIONS:
Overall Officials: Gilles Rode, PhD, Study Chair — Claude Bernard University; Marc Lilot, PhD, Study Director — Claude Bernard University
Locations (1):
- Claude Bernard University, Lyon, France

IPD SHARING:
Plan to Share IPD: No
Protocol will be available on request